CLINICAL TRIAL: NCT04224493
Title: Symphony-1: A Phase 1b/3 Double-Blind, Randomized, Active-Controlled, 3-Stage, Biomarker Adaptive Study Of Tazemetostat Or Placebo In Combination With Lenalidomide Plus Rituximab In Subjects With Relapsed/Refractory Follicular Lymphoma
Brief Title: A Study to Assess the Efficacy, Safety, Pharmacodynamics, and Pharmacokinetics of Tazemetostat in Combination With Lenalidomide Plus Rituximab Versus Placebo in Combination With Lenalidomide Plus Rituximab in Adult Patients at Least 18 Years of Age With Relapsed/Refractory Follicular Lymphoma.
Acronym: SYMPHONY-1
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EZH-302; 2019-003333-42 (EudraCT Number); 2024-510690-16-00 (EU CTIS Number)
Record Dates: First submitted 2019-12-12; First posted 2020-01-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Relapsed/Refractory Follicular Lymphoma; Follicular Lymphoma; Refractory Follicular Lymphoma
Keywords: Epizyme; Tazverik; Tazemetostat (EPZ-6438); Lenalidomide; Revlimid; Rituximab; Rituxan; Follicular lymphoma; EZH2
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tazemetostat; Lenalidomide; Rituximab

STUDY DESIGN:
Intervention Model Description: 3 stages study:
  Stage 1:
  Open-Label (Phase 1b: Safety run-in): All participants will receive Tazemetostat in combination with Lenalidomide and Rituximab
  Stage 2:
  Double-blinded (Phase 3):
  * Study drug arm: Tazemetostat in combination with Lenalidomide and Rituximab
  * Placebo arm: Placebo in combination with Lenalidomide and Rituximab
  Stage 3:
  Long-term Follow-up of participants in Stage 2 after treatment for response, when applicable, and overall survival for up to 5 years after the enrollment of the last patient in the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tazemetostat + R2 arm (Experimental): Stage 1 (Phase 1b): This phase is now completed.
  * Tazemetostat was escalated from a starting dose of 400 mg PO twice daily to 600 mg PO twice daily to 800 mg PO twice daily in 28-day cycles.
  * Rituximab 375 mg/m2 IV on days 1, 8, 15, and 22 of cycle 1; then on day 1 of cycles 2 to 5.
  * Lenalidomide 20 mg or 10 mg (if creatinine clearance ≥60 mL/minute or <60 mL/minute), administred PO QD on days 1 to 21 for 12 cycles.
  Stage 2:
  * Tazemetostat 800 mg administered PO twice daily in continuous 28-day cycles.
  * Rituximab 375 mg/m2 IV on days 1, 8, 15, and 22 of cycle 1; then on day 1 of cycles 2 to 5.
  * Lenalidomide 20 mg or 10 mg (if creatinine clearance ≥60 mL/minute or <60 mL/minute), PO QD on days 1 to 21 for 12 cycles.
  Maintenance Therapy (Stages 1 and 2):
  Tazemetostat will be administered as monotherapy at an 800 mg twice daily dose for up to 2 years after the initial 12 months of combination therapy.
  Interventions: Drug: Tazemetostat; Combination Product: Lenalidomide; Combination Product: Rituximab
- Placebo + R2 Arm (Placebo Comparator): Stage 2:
  * Placebo administered PO twice daily in continuous 28-day cycles.
  * Rituximab 375 mg/m2 IV on days 1, 8, 15, and 22 of cycle 1; then on day 1 of cycles 2 to 5.
  * Lenalidomide 20 mg or 10 mg (if creatinine clearance ≥60 mL/minute or <60 mL/minute), administered PO QD on days 1 to 21 for 12 cycles.
  Maintenance Therapy (Stage 2):
  Placebo will be administered as monotherapy twice daily dose for up to 2 years after the initial 12 months of combination therapy. During maintenance, placebo will be continued until disease progression or unacceptable toxicity, or participant withdraws consent.
  Interventions: Drug: Placebo oral tablet; Combination Product: Lenalidomide; Combination Product: Rituximab

INTERVENTIONS:
Drug: Tazemetostat — Stage 1 (Phase 1b):
  Tazemetostat was escalated from a starting dose of 400 mg orally twice daily to 600 mg orally twice daily to 800 mg PO twice daily in 28-day cycles as tolerated in a standard 3 + 3 design. Tazemetostat will be administered as monotherapy at an 800 mg twice daily dose for up to 2 years after the initial 12 months of combination therapy.
  Other Names: EPZ-6438; IPN60200
  Arms: Tazemetostat + R2 arm
Drug: Tazemetostat — Stage 2:
  Tazemetostat 800 mg administered orally twice daily in continuous 28-day cycles for 12 cycles. Tazemetostat will be administered as monotherapy at an 800 mg twice daily dose for up to 2 years after the initial 12 months of combination therapy.
  Other Names: EPZ-6438; IPN60200
  Arms: Tazemetostat + R2 arm
Drug: Placebo oral tablet — Stage 2:
  Placebo administered orally twice daily in continuous 28-day cycles. Placebo will be administered as monotherapy twice daily dose for up to 2 years after the initial 12 months of combination therapy.
  Arms: Placebo + R2 Arm
Combination Product: Lenalidomide — Lenalidomide 20 mg capsules or 10 mg capsules (if creatinine clearance ≥60 mL/minute or <60 mL/minute), administered PO QD on days 1 to 21 for 12 cycles.
Combination Product: Rituximab — Rituximab 375 mg/m2 IV on days 1, 8, 15, and 22 of cycle 1; then on day 1 of cycles 2 to 5.

SUMMARY:
The participants of this study would have relapsed/refractory follicular lymphoma.

Follicular lymphoma is a type of blood cancer. It is referred to as 'relapsed' when the disease has come back after a period of improvement after that follows a treatment regimen and 'refractory' when treatment no longer works.

Stage 1 of this trial will study the safety and the level that adverse effects of each of the study drug combinations can be tolerated (known as tolerability). It is also designed to establish a recommended study drug dosage for stage 2 and 3. Stage 1 of the study is completed.

Stages 2 and 3 will evaluate and compare how long participants live without their disease getting worse when receiving the study drug in combination with other drug treatment versus the placebo (dummy drug) in combination with other drug treatment.

DETAILED DESCRIPTION:
Stage 1 of the study, which is now completed, looked at the safety and tolerability of the drug combinations and helped determine the recommended dose for the next stages.

In Stage 2, participants will be grouped based on whether they have a specific genetic mutation called EZH2. All participants will receive treatment in 28-day cycles. After 12 cycles, they will continue with maintenance treatment using either the study drug or a placebo, depending on their original group.

The study will include participants with and without the EZH2 mutation. Enrollment may be completed separately for each group. In China, some participants will also have extra blood tests to better understand how the drug behaves in the body.

Stage 3 will focus on long-term follow-up to monitor how well the treatment works, how safe it is, and how long participants live. All participants will be followed for up to 5 years after the last person joins the study

ELIGIBILITY:
Inclusion Criteria:

1. Have voluntarily agreed to provide written informed consent and demonstrated willingness and ability to comply with all aspects of the protocol.
2. Males or females are ≥18 years of age, or per country adult legal age regulations, at the time of providing voluntary written informed consent.
3. Life expectancy ≥3 months before enrollment.
4. Meet requirement for hepatitis and human immunodeficiency virus (HIV) infection as follows

   * Negative serologic or polymerase chain reaction (PCR) test results for acute or chronic hepatitis B virus (HBV) infection Note: Participants whose HBV infection status could not be determined by serologic test results have to be negative for HBV-DNA by PCR to be eligible for study participation. Participants seropositive for HBV with undetectable HBV DNA by PCR are permitted with appropriate antiviral prophylaxis.
   * Negative test results for hepatitis C virus (HCV) Note: Participants who are positive for HCV antibody must be negative for HCV RNA by PCR to be eligible for study participation
   * If HIV positive, HIV infection is controlled. Based on Cancer Clinical Trial Eligibility Criteria: Patients with HIV, Hepatitis B Virus, or Hepatitis C Virus Infections - Guidance for Industry (https://www.fda.gov/media/121319/download), patients with HIV should be considered eligible if they have CD4+ T-cell counts ≥ 350 cells/uL and in general, if they have not had an opportunistic infection within the past 12 months. Other exclusion criteria should be considered regarding the drug-drug interaction if antiviral drugs are used. Therefore, in case of controlled HIV infection, since antiviral drugs are used, trial patients should be on established ART for at least 4 weeks and have an HIV viral load less than 400 copies/mL prior to enrolment.
5. Have histologically confirmed FL, Grades 1 to 3A.
6. Must have been previously treated with at least 1 prior systemic chemotherapy, immunotherapy, or chemoimmunotherapy:

   a. Systemic therapy includes treatments such as:

   i. Rituximab monotherapy

   ii. Chemotherapy given with or without rituximab

   iii. Radioimmunoconjugates such as 90Y-ibritumomab tiuxetan and 131I-tositumomab.

   b. Systemic therapy does not include, for example:

   i. Local involved field radiotherapy for limited-stage disease

   ii. Helicobacter pylori eradication

   c. Prior investigational therapies will be allowed provided the subject has received at least 1 prior systemic therapy as discussed in Inclusion Criterion #6a.

   d. Prior autologous/allogeneic hematopoietic stem cell transplant (HSCT) will be allowed.

   e. Prior chimeric antigen receptor T-cell therapy (CAR T) will be allowed.
7. Must have documented relapsed, refractory, or PD after treatment with systemic therapy (refractory defined as less than PR or disease progression <6 months after last dose).
8. Have measurable disease as defined by the Lugano Classification (Cheson, 2014; Appendix 5).
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
10. Within 7 days prior to randomization, all clinically significant toxicity related to a prior anticancer treatment (ie, chemotherapy, immunotherapy, and/or radiotherapy must have either resolved to Grade 1 per NCI CTCAE Version 5.0 OR are clinically stable and no longer clinically significant.
11. Have provided sufficient tumor tissue block or unstained slides for EZH2 mutation testing in all subjects to allow for stratification

    a. If EZH2 mutation status is known from site-specific testing, subjects can be enrolled. Tumor tissue will be required for confirmatory testing of EZH2 status at study-specific laboratories. If the archival tumor sample was collected more than 24 months prior to the anticipated administration of the first dose (cycle 1 day 1), then a fresh biopsy must be provided. Fresh tumor biopsy is appropriate except for procedures deemed to result in unacceptable risk because of the anatomical location including brain, lung/mediastinum, pancreas, or endoscopic procedures extending beyond the esophagus, stomach, or bowel. Archival tumor biopsy sections mounted on slides are also acceptable.

    NOTE: Confirmatory testing will also be performed for Stage 1, if local EZH2 testing is conducted, unless there is insufficient tumor tissue to perform testing after discussion with the Sponsor's or Designee Medical Monitor.
12. Time between prior anticancer therapy and first dose of tazemetostat as follows:

    1. Cytotoxic chemotherapy - At least 21 days.
    2. Noncytotoxic chemotherapy (eg, small molecule inhibitor) - At least 14 days.
    3. Nitrosoureas - At least 6 weeks.
    4. Monoclonal and/or bispecific antibodies or CAR T - At least 28 days.
    5. Radiotherapy - At least 6 weeks from prior radioisotope therapy; at least 12 weeks from 50% pelvic or total body irradiation.
13. Adequate renal function defined as calculated creatinine clearance ≥30 mL/minute per the Cockcroft and Gault formula.
14. Adequate bone marrow function:

    a. Absolute neutrophil count (ANC) ≥1000/mm3 (≥1.0 × 10^9/L) if no lymphoma infiltration of bone marrow OR ANC ≥750/mm3 (≥75 × 10^9/L) with bone marrow infiltration
    * Without growth factor support (filgrastim or pegfilgrastim) for at least 14 days.

      b. Platelets ≥75,000/mm3 (≥75 × 10^9/L)
    * Evaluated at least 7 days after last platelet transfusion.

      c. Hemoglobin ≥9.0 g/dL
    * May receive transfusion
15. Adequate liver function:

    1. Total bilirubin ≤1.5 × the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome.
    2. Alkaline phosphatase (ALP) (in the absence of bone disease), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤3 × ULN (≤5 × ULN if subject has liver infilration).
16. International normalized ratio (INR) ≤1.5 × ULN and activated partial thromboplastin time (aPTT) ≤1.5 × ULN (unless on warfarin, then INR ≤3.0). In subjects with thromboembolism risk, prophylactic anticoagulation, or antiplatelet therapy at investigator discretion is recommended.
17. Females of childbearing potential (FCBP) must have a negative urine or serum pregnancy tests (beta-human chorionic gonadotropin [β-hCG] tests with a minimum sensitivity of 25 mIU/mL or equivalent units of β-hCG) at screening within 10 to 14 days prior to first dose of study drug. The subject may not receive study drug until the study doctor has verified that the results of pregnancy tests are negative. All females will be considered to be of childbearing potential unless they are naturally postmenopausal (at least 24 months consecutively amenorrhoeic [amenorrhea following cancer therapy does not rule out childbearing potential] and without other known or suspected cause) or have been sterilized surgically (ie, total hysterectomy and/or bilateral oophorectomy, with surgery completed at least 1 month before dosing).
18. Females of childbearing potential (FCBP) enrolled must either practice complete abstinence or agree to use two reliable methods of contraception simultaneously. This includes ONE highly effective method of contraception and ONE additional effective contraceptive method. Contraception must begin at least 28 days prior to first dose of study drug, continue during study treatment (including during dose interruptions), and for 12 months after study drug discontinuation. Female subjects must also refrain from breastfeeding for 12 months following last dose of study drug. If the below contraception methods are not appropriate for the FCBP, she must be referred to a qualified contraception provider to determine the medically effective contraception method appropriate for the subject. The following are examples of highly effective and additional effective methods of contraception:

    Examples of highly effective methods:
    * Intrauterine device (IUD)
    * Hormonal (ovulation inhibitory combined [estrogen and progesterone] birth control pills or intravaginal/transdermal system, injections, implants, levonorgestrel-releasing intrauterine system [IUS], medroxyprogesterone acetate depot injections, ovulation inhibitory progesterone-only pills [e.g. desogestrel]) NOTE: There is a potential for tazemetostat interference with hormonal contraception methods due to enzymatic induction.
    * Bilateral tubal ligation
    * Partner's vasectomy (if medically confirmed [azoospermia] and sole sexual partner).

    Examples of additional effective methods:
    * Male latex or synthetic condom,
    * Diaphragm,
    * Cervical Cap

    NOTE: Female subjects of childbearing potential exempt from these contraception requirements are subjects who practice complete abstinence from heterosexual sexual contact. True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, or post ovulation methods) and withdrawal are not acceptable methods of contraception.
19. All study participants enrolled must be registered into the applicable pregnancy prevention program (e.g. REVLIMID REMS in the US, Pregnancy Prevention Programme [PPP] in Europe) for lenalidomide to be administered and be willing and able to comply with the requirements of the applicable program as appropriate for the country in which the drug is being used.

    a. Female subjects of childbearing potential (FCBP) must adhere to the scheduled pregnancy testing as required in theapplicable pregnancy prevention program. During study treatment, FCBP must agree to have pregnancy testing weekly for the first 28 days of study participation and then every 28 days for FCBP with regular or no menstrual cycles OR every 14 days for FCBP with irregular menstrual cycles. FCBP must also have a pregnancy test at end of lenalidomide treatment, at day 14 (for FCBP with irregular menstrual cycles) and day 28 following the last dose of lenalidomide and at overall treatment discontinuation (at the End-of-Treatment/30-day safety Follow-up visit). Female subjects exempt from this requirement are subjects who have been naturally postmenopausal for at least 24 consecutive months OR are surgically sterilized (ie, total hysterectomy or bilateral oophorectomy) with surgery at least 1 month before the first dose of study treatment.
20. Male subjects must either practice complete abstinence or agree to use a latex or synthetic condom, even with a successful vasectomy (medically confirmed azoospermia), during sexual contact with a pregnant female or FCBP from first dose of study drug, during study treatment (including during dose interruptions), and for 3 months after study drug discontinuation.

NOTE: Male subjects must not donate semen or sperm from first dose of study drug, during study treatment (including during dose interruptions), and for 3 months after study drug discontinuation.

Exclusion Criteria:

All Subjects

1. Prior exposure to tazemetostat or other inhibitor(s) of EZH2.
2. Prior exposure to lenalidomide or drugs of the same class.
3. Grade 3b, mixed histology, or FL that has histologically transformed to diffuse large B-cell lymphoma (DLBCL) (subjects transformed from DLBCL to FL may be enrolled).
4. Has thrombocytopenia, neutropenia, or anemia of Grade ≥3 (per CTCAE Version 5.0 criteria) or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or myeloproliferative neoplasm (MPN).
5. Has a prior history of T-cell lymphoblastic lymphoma (T-LBL)/T-cell acute lymphoblastic leukemia (T-ALL) or B-cell acute lymphoblastic leukemia (B-ALL).
6. Subjects with uncontrolled leptomeningeal metastases or brain metastases or history of previously treated brain metastases.
7. Subjects taking medications that are known strong CYP3A inhibitors and strong or moderate CYP3A inducers (including St. John's wort).
8. Are unwilling to exclude grapefruit juice, Seville oranges, and grapefruits from the diet and/or consumed within 1 week of the first dose of study drug and for the duration of the study.
9. Major surgery within 4 weeks before the first dose of study drug.

   a. Note: Minor surgery (eg, minor biopsy of extracranial site, central venous catheter placement, shunt revision) is permitted within 3 weeks prior to enrollment.
10. Are unable to take oral medication OR have malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, vomiting) that might impair the bioavailability of tazemetostat.
11. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac ventricular arrhythmia.
12. Prolongation of corrected QT interval using Fridericia's formula (QTcF) to ≥480 msec at screening or history of long QT syndrome.
13. Venous thrombosis or pulmonary embolism within the last 3 months before starting tazemetostat.

    a. Note: Participants who have experienced deep vein thrombosis/pulmonary embolism more than 3 months before enrollment are eligible but are recommended to receive prophylaxis.
14. Have an active infection requiring systemic therapy.
15. Known hypersensitivity to any component of tazemetostat or lenalidomide; known severe hypersensitivity to any component of rituximab requiring hospitalization or resuscitation.
16. Active viral infection with or seropositive for HBV: HBV surface antigen (HBsAg) positive OR HBsAg negative, anti-HBs positive and/or anti-HBc positive with detectable HBV DNA.

    NOTE: Subjects who are HBsAg negative, anti-HBs positive and/or anti-HBc positive, but with undetectable viral DNA and normal ALT are eligible. Subjects who are seropositive due to HBV vaccination (HBsAg negative, HBV surface antibody [anti-HBs] positive, and HBV core antibody [anti-HBc] negative) are eligible.
17. Active viral infection with hepatitis C virus (as measured by positive HCV antibody and detectable viral RNA, HIV), or known active infection with human T-cell lymphotropic virus.

    NOTE: Subjects with a history of hepatitis C infection (HCV antibody reactive) who have normal ALT and undetectable HCV RNA are eligible.
18. Any other medical or social condition that, in the Investigator's judgment, will interfere with a participant's ability to provide informed consent, to receive study drugs, or meet study demands, or that substantially increases the risk associated with the subject's participation in the study, or that may interfere with interpretation of results.
19. Female subjects who are pregnant or lactating/breastfeeding.
20. Subjects who have undergone a solid organ transplant.
21. Subjects with malignancies other than FL. a. Exception: Subjects with another malignancy who have been disease-free for 3 years, or subjects with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 612 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 3 Dose (RP3D) of tazemetostat in combination with rituximab and lenalidomide (R2) | Subjects are evaluated for DLTs during the first 28-day cycle. The RP3D for Phase 3 was selected at the end of Stage 1
  The safety and tolerability of tazemetostat in combination with R2 in subjects with R/R FL will be evaluated. RP3D of tazemetostat for further evaluation in phase 3 will be selected as assessed by the occurrence of treatment-emergent dose-limiting toxicities (DLTs) and adverse events (AEs).
Progression-Free Survival (PFS) in the Intent-to-treat wild-type (ITT-WT) population | Stage 2: Up to 72 months
  PFS is defined as the time from the date of randomization to the time of confirmed disease progression per the 2014 Lugano Classification or death, whichever occurs first, as assessed by Investigators.
PFS in the Intent-to-treat mutant-type (ITT-MT) population | Stage 2: Up to 72 months
  PFS is defined as the time from the date of randomization to the time of confirmed disease progression per the 2014 Lugano Classification or death, whichever occurs first, as assessed by Investigators.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of tazemetostat: Maximum (peak) Observed Plasma Drug Concentration (Cmax). | Stage 1: In cycles 1 and 2 on days 1 and 15 (28 days cycle)
  Cmax will be recorded from the PK blood samples collected.
PK of tazemetostat, EPZ 6930 (desethyl metabolite), and lenalidomide as data permit: Time to Maximum Observed Drug Concentration (Tmax) | Stage 1: In cycles 1 and 2 on days 1 and 15 (28 days cycle)
PK of tazemetostat: area under the plasma concentration-time curve (AUC) from time 0 to the time of the last quantifiable concentration [AUC(0-t)], | Stage 1: In cycles 1 and 2 on days 1 and 15 (28 days cycle)
PK of tazemetostat: area under the plasma concentration-time curve (AUC) from time 0 to infinity [AUC(0-∞)] | Stage 1: In cycles 1 and 2 on days 1 and 15 (28 days cycle)
The apparent terminal elimination half-life (t1/2) of tazemetostat, EPZ 6930 (desethyl metabolite), and lenalidomide as data permit | Stage 1: In cycles 1 and 2 on days 1 and 15 (28 days cycle)
Complete Response Rate (CRR) in ITT-WT population | Stage 2: Up to 96 months
  CRR is defined as the proportion of participants achieving CR according to the 2014 Lugano Classification, as assessed by the Investigator and a blinded Independent Review Committee (IRC).
CRR in ITT-MT population | Stage 2: Up to 96 months
  CRR is defined as the proportion of participants achieving CR according to the 2014 Lugano Classification, as assessed by the Investigator and a blinded IRC.
CRR in the Relapsed/Refractory (R/R) Follicular Lymphoma (FL) population regardless of mutation status | Stage 2: Up to 96 months
  CRR is defined as the proportion of participants achieving CR according to the 2014 Lugano Classification, as assessed by the Investigator and a blinded IRC.
Objective Response Rate (ORR) in the ITT-WT population | Stage 2: Up to 96 months
  ORR is defined as the proportion of participants achieving a best overall response (BOR) of partial response (PR) or complete response (CR) according to the 2014 Lugano Classification, as assessed by the Investigator and a blinded IRC.
ORR in the ITT-MT population | Stage 2: Up to 96 months
  ORR is defined as the proportion of participants achieving a best overall response (BOR) of partial response (PR) or complete response (CR) according to the 2014 Lugano Classification, as assessed by the Investigator and a blinded IRC.
ORR in the R/R FL population regardless of mutation status | Stage 2: Up to 96 months
  ORR is defined as the proportion of participants achieving a best overall response (BOR) of partial response (PR) or complete response (CR) according to the 2014 Lugano Classification, as assessed by the Investigator and a blinded IRC.
Overall Survival (OS) in the ITT-WT population | Stage 2: Up to 96 months
  OS is defined as the time from the date of randomization until death due to any cause.
OS in the ITT-MT population | Stage 2: Up to 96 months
OS in the R/R FL population regardless of mutation status | Stage 2: Up to 96 months
PFS in the ITT-WT population, assessed by a blinded IRC | Stage 2: Up to 96 months
PFS in the ITT-MT population, assessed by a blinded IRC | Stage 2: Up to 96 months
PFS in the R/R FL population regardless of mutation status, assessed by a blinded IRC | Stage 2: Up to 96 months
PFS in the R/R FL population regardless of mutation status, assessed by the Investigator | Stage 2: Up to 96 months
Duration Of Response (DOR) in the ITT-WT population | Stage 2: Up to 96 months
  DOR is defined as the time from initial CR or PR to documented progression or death due to any cause, whichever occurs first, for those participants with a CR or PR, as assessed by the Investigator and by a blinded IRC.
DOR in the ITT-MT population | Stage 2: Up to 96 months
  DOR is defined as the time from initial CR or PR to documented progression or death due to any cause, whichever occurs first, for those participants with a CR or PR, as assessed by the Investigator and by a blinded IRC.
DOR in the R/R FL population regardless of mutation status | Stage 2: Up to 96 months
  DOR is defined as the time from initial CR or PR to documented progression or death due to any cause, whichever occurs first, for those participants with a CR or PR, as assessed by the Investigator and by a blinded IRC.
Duration Of Complete Response (DOCR) in the ITT-WT population | Stage 2: Up to 96 months
  DOCR is defined as the time from initial CR to documented progression or death due to any cause, whichever occurs first, for those participants with CR, assessed by the Investigator and by a blinded IRC.
DOCR in the ITT-MT population | Stage 2: Up to 96 months
  DOCR is defined as the time from initial CR to documented progression or death due to any cause, whichever occurs first, for those participants with CR, assessed by the Investigator and by a blinded IRC.
DOCR in the R/R FL population regardless of mutation status | Stage 2: Up to 96 months
  DOCR is defined as the time from initial CR to documented progression or death due to any cause, whichever occurs first, for those participants with CR, assessed by the Investigator and by a blinded IRC.
Disease Control Rate (DCR) in the ITT-WT population | Stage 2: Up to 96 months
  DCR, defined as the proportion of participants with best overall response of CR, PR, or stable disease (SD) lasting 12 or more months, as assessed by the Investigator and by a blinded IRC.
DCR in the ITT-MT population | Stage 2: Up to 96 months
  DCR, defined as the proportion of participants with best overall response of CR, PR, or stable disease (SD) lasting 12 or more months, as assessed by the Investigator and by a blinded IRC.
DCR in the R/R FL population regardless of mutation status | Stage 2: Up to 96 months
  DCR, defined as the proportion of participants with best overall response of CR, PR, or stable disease (SD) lasting 12 or more months, as assessed by the Investigator and by a blinded IRC.
Population PK parameters of oral clearance (CL/F) of tazemetostat | Stage 2: In cycles 2, 4, 6, and 12 at Day 1 (28 days cycle)
  CL/F will be used to generate estimates of tazemetostat AUC
Population PK parameters of oral volume of distribution (Vd/F) of tazemetostat. | Stage 2: In cycles 2, 4, 6, and 12 at Day 1 (28 days cycle)
Population PK parameters of first-order absorption rate constant (Ka) for tazemetostat. | Stage 2: In cycles 2, 4, 6, and 12 at Day 1 (28 days cycle)
Percentage of Participants Experiencing Adverse Events (AEs) | Up to 36 months
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Percentage of Participants with Clinically Significant Changes in Physical Examination | Up to 36 months
  Percentage of participants with clinically significant changes in physical examination findings will be reported. The clinical significance will be graded by the investigator according to the National Cancer Institute Common Terminology Criteria for AEs (CTCAE) Version 5.0.
Percentage of Participants with Clinically Significant Changes in Vital Signs | Up to 36 months
  Percentage of participants with clinically significant changes in vital signs findings will be reported. The clinical significance will be graded by the investigator according to the National Cancer Institute Common Terminology Criteria for AEs (CTCAE) Version 5.0.
Percentage of Participants with Clinically Significant Changes in Electrocardiogram (ECG) Readings | Up to 72 months
  Percentage of participants with clinically significant changes in ECG Readings will be reported. The clinical significance will be graded by the investigator according to the National Cancer Institute Common Terminology Criteria for AEs (CTCAE) Version 5.0.
Performance status evaluated by Eastern Cooperation Oncology Group (ECOG) | Up to 72 months
  ECOG is a 6-point performance status scale used to assess performance using PA as a key indicator (e.g., 0 = fully active, 2 = up and about more than 50% of walking hours, 5 = dead) Performance status will be assessed per usual clinical practice and will be recorded in the medical record.
Duration of Study Drug Exposure | Up to 36 months
  Duration of exposure to study drug will be reported.
Percentage of study drug taken by participants | Up to 36 months
Quality of life questionnaires evaluation | Up to 36 months
  Evaluate and compare health-related quality of life as measured by the EuroQOL 5-Dimension 5-Level (EQ-5D-5L) instrument and the Functional Assessment of Cancer Therapy -Lymphoma (FACT-Lym)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (229):
- United States (77):
  - Southern Cancer Center, Mobile, Alabama
  - Arizona Oncology Associates - Tuscon-Rusadill Road, Tucson, Arizona
  - TOI - Clinical Research, Cerritos, California
  - UCSF Fresno, Clovis, California
  - UC San Diego Health Sciences, La Jolla, California
  - UCLA Clinical Research Unit Hematology/Oncology, Santa Monica, California
  - Rocky Mountain Cancer Centers (RMCC) - Boulder, Boulder, Colorado
  - St. Mary's Hospital and Regional Medical Center - St. Mary's, Grand Junction, Colorado
  - SCL Health Lutheran Medical Center, Greeley, Colorado
  - Cancer Specialists of North Florida, Fleming Island, Florida
  - Florida Cancer Specialists & Research Institute (FCS) - Fort Myers Cancer Center, Fort Myers, Florida
  - Mayo Clinic - Cancer Clinical Research Office, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Florida Cancer Affiliates/Ocala Oncology - Clinic, Ocala, Florida
  - BRCR Medical Center, INC, Plantation, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists - Panhandle, Tallahassee, Florida
  - H Lee Moffitt Cancer Center and Research Institute I, Tampa, Florida
  - Florida Cancer Specialists & Research Institute (FCS) - Atlantis, West Palm Beach, Florida
  - Kaiser Permanente Hawaii Moanalua Medical Center, Honolulu, Hawaii
  - University of Chicago, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - June E. Nylen Cancer Center, Sioux City, Iowa
  - The University of Kansas Cancer Center, Overland Park, Kansas
  - University of Maryland, Baltimore, Maryland
  - The office of Frederick P. Smith, MD, P.C., Chevy Chase, Maryland
  - Mass General Cancer Center at Newton-Wellesley, Newton, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Saint Louis University Cancer Center, St Louis, Missouri
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Astera Cancer Care, East Brunswick, New Jersey
  - Astera Cancer Center, East Brunswick, New Jersey
  - Regional Cancer Care Associates-Freehold, Freehold, New Jersey
  - Hackensack University Medical John Theurer Cancer Center, Hackensack, New Jersey
  - Regional Cancer Care Associates LLC - Howell, Howell Township, New Jersey
  - Regional Cancer Care Associates LLC - Little Silver, Little Silver, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - New York Oncology Hematology, P.C., Albany, New York
  - Northwell Health/Monter Cancer Center, Lake Success, New York
  - Weill Cornell Medicine-New York Presbyterian Hospital, New York, New York
  - Columbia U - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Hematology Oncology Associates of Rockland, P.C., Nyack, New York
  - Messino Cancer Center, Asheville, North Carolina
  - Levine Cancer Institute - Concord, Concord, North Carolina
  - FirstHealth of the Carolinas, Pinehurst, North Carolina
  - Regional Medical Oncology Center, Wilson, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Oncology Hematology Care (OHC), Inc. - Kenwood Office, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center - Oncology, Eugene, Oregon
  - University of Pittsburgh Medical Center - Oncology, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital Hematology & Cellular Therapy, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC, Chattanooga, Tennessee
  - University of Tennessee Medical Center - Cancer Institute, Knoxville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Medical City Dallas Pediatric Hematology, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Millennium Physicians - Oncology, Houston, Texas
  - Texas Oncology, Plano, Texas
  - Mays Cancer Center, San Antonio, Texas
  - UT Health East Texas HOPE Cancer Center - Tyler, Tyler, Texas
  - USO Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology- Weslaco, Weslaco, Texas
  - Utah Cancer Specialists/ IHO Corp, Salt Lake City, Utah
  - Huntsman Cancer Institute; The University of Utah, Salt Lake City, Utah
  - Peninsula Cancer Institute, Chesapeake, Virginia
  - Virginia Cancer Specialists, Gainesville, Virginia
  - Oncology and Hematology Associates of Southwest Virginia Inc., Roanoke, Virginia
  - MC Rockwood Cancer Bl Specialty Ctr - North, Spokane, Washington
  - Yakima Valley Memorial Hospital - North Star Lodge Cancer Center, Yakima, Washington
  - Wheeling Hospital, Wheeling, West Virginia
- Australia (9):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Health, Clayton, Victoria
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - Hollywood Private Hospital, Nedlands, Western Australia
  - GenesisCare - St Andrew's, Adelaide
  - Peninsula Health - Frankston, Frankston
  - Royal Hobart Hospital, Hobart
  - Gold Coast University Hosptial, Southport
- Belgium (3):
  - CHU Dinant Godinne UCL Namur, Yvoir, Namur
  - Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven - Campus Gasthuisberg, Leuven, Vlaams Brabant
- Brazil (14):
  - Hospital Haroldo Juacaba - Instituto do Cancer do Ceara, Ceará
  - Hospital Santa Cruz, Curitiba
  - HC-UFG - Hospital das CLINICAS da Universidade Federal de Go, Goiânia
  - Association Hospital de Caridade de Iju, Ijuí
  - Liga Norte Riograndense Contra o Cancer, Natal
  - Hospital de Clinicas de Porto Alegre - Centro de Pesquisa Clinica, Porto Alegre
  - Instituto D'Or de Pesquisa e Ensino- Recife, Recife
  - Instituto de Psiquiatria - UFRJ, Rio de Janeiro
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
  - Fundacao Antonio Prudente - Hospital A.C.Camargo Cancer Center, São Paulo
  - Hospital Alemao Oswaldo Cruz (HAOC), São Paulo
  - Instituto D'or de Pesquisa e Ensino, São Paulo
  - Instituto de Oncologia e Hematologia - HEMOMED, São Paulo
  - Irmandade Santa Casa de Misericordia de Sao Paulo, São Paulo
- Canada (5):
  - University Health Network Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - Sir Mortimer B Davis/Jewish General Hospital, Montreal, Quebec
  - Nova Scotia Health Centre for Clinical Research, Nova Scotia
  - Sunnybrook Health Sciences Centre Odette Cancer Centre, Ottawa
- China (20):
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Zhejiang, Hangzhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Bethune Hospital of Jilin University, Changchun, Jinlin
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Peking University Third Hospital, Beijing
  - The First Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Tongji Hospital of Tongji Medical College of HUST, Hangzhou
  - Jiangxi Cancer Hospital, Nanchang
  - Shandong Cancer Hospital, Shandong
  - Tongji Hospital of Tongji University, Shanghai
  - Sichuan Provincial People's Hospital, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
- France (24):
  - Centre Hospitalier Universitaire de Bordeaux-Hopital du Haut Leveque, Pessac, Aquitaine
  - CHRU Brest Hôp Morvan, Brest, Brittany Region
  - Institut Bergonie, Bordeaux, Gironde
  - Centre Hosp Mulh Hop Emile Muller, Mulhouse, Haut-Rhin
  - Centre Henri Becquerel, Rouen, Haute-Normandie
  - CHU de Limoges Dupuytren, Limoges, Haute-Vienne
  - CHU de Grenoble - Hopital Albe, La Tronche, Isere
  - CHU de Nantes - Hematologie, Nantes, Loire-Atlantique
  - CHRU de Lille Hop Claude Huriez, Lille, Nord
  - Centre Hospitalier Le Mans, Le Mans, Sarthe
  - Centre Hospitalier Universitaire D'Angers - Hématologie Clinique, Angers
  - CHRU de Besançon- Hopital Jean Minjoz, Besançon
  - CHU Caen, Caen
  - CHU de Clermont-Ferrand, site Estaing, Clermont-Ferrand
  - Centre Hospitalier Docteur Schaffner, Lens
  - L'Hôpital Privé Confluent, Nantes
  - L'hôpital Privé du Concluent, Nantes
  - Hopital Saint Louis, Paris
  - Centre Hospitalier - Hôpital de jour d'Hématologie, Périgueux
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - CHU de Nancy Brabois, Vandœuvre-lès-Nancy
  - Centre Hospitalier Bretagne Atlantique, Vannes
  - Institut Gustave Roussy, Villejuif
  - Hopital Henri Mondor - Hemopathies Lymphoides, Créteil, Île-de-France Region
- Germany (9):
  - Diakoneo Diak Schwaebisch Hall gGmbH, Schwäbisch Hall, Baden-Wurttemberg
  - Klinikum Der Universität München AöR, München, Bavaria
  - Klinikum rechts der Isar der Technischen Universitat Muenche, München, Bavaria
  - Universitätsmedizin Mainz, Mainz, Hesse
  - Universitaetsklinikum Bonn AöR, Bonn, North Rhine-Westphalia
  - Kliniken Maria Hilf GmbH, Mönchengladbach, North Rhine-Westphalia
  - Städt. Krankenhaus Kiel, Kiel, Schleswig-Holstein
  - Vivantes Klinikum am Urban Hämatologie und Onkologie, Berlin
  - University Medical Center Schleswig Holstein, Kiel
- Hungary (4):
  - Debreceni Egyetem Klinikai Központ, Debrecen, Hajdú-Bihar
  - Semmelweis Egyetem Általános Orvostudományi Kar, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Del-pesti Centrumkorhaz Orszagos Hematologiai és Infektologiai Intezet, Budapest
- Italy (19):
  - AOU Federico II, Napoli, Campania
  - Istituto Romagnolo per lo Studio dei Tumori (IRST) Dino Amadori IRCCS, Meldola, Forli-Cesena
  - ASST Spedali Civili di Brescia, Brescia
  - PO Garibaldi-Nesima, ARNAS Garibaldi, Catania
  - AOU Careggi, Florence
  - Ospedale Vito Fazzi, ASL Lecce, Lecce
  - IEO - Istituto Europeo di Oncologia, IRCCS, Milan
  - Ospedale Maggiore Policlinico, Fondazione IRCCS Ca' Granda, Milan
  - Ospedale Niguarda, ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Ospedale San Gerardo, ASST di Monza, Monza
  - Ospedale Civile S.Spirito, PO di Pescara, AUSL Pescara, Pescara
  - Ospedale Infermi di Rimini, AUSL Rimini, Distretto di Rimini, Presidio di Rimini, Santarcangelo di Romagna e Novafeltria, Rimini
  - Catholic University Of Sacred Heart, Roma
  - PU Campus Bio-Medico di Roma, Roma
  - Regina Elena, Istituto Nazionale dei Tumori , IFO, IRCCS, Roma
  - Azienda Ospedaliera Santa Maria di Terni, Terni
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Ospedale Umberto I di Torino, Torino
  - Ospedale S.Giacomo Apostolo, PO Castelfranco Veneto, AULSS 2 Marca Trevigiana, Treviso
  - Azienda Sanitaria Universitaria Giuliano Isontina (ASU GI), Ospedale Maggiore, Trieste
- Poland (8):
  - Centrum Medyczne Pratia Poznan, Skórzewo, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Pratia Onkologia Katowice, Katowice
  - Pratia MCM Krakow, Krakow
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Slupsku Sp. z o.o., Słupsk
  - MICS Centrum Medyczne Torun, Torun
  - MTZ Clinical Research powered by Pratia, Warsaw
  - Uniwersytecki Szpital Kliniczny im. J. Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Singapore (2):
  - National Cancer Center Singapore, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (7):
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Pusan National University Hospital, Busan
  - Gachon University Gil Medical Center, Incheon
  - Ajou University Hospital, Suwon
- Spain (11):
  - Hospital Universitari Vall d'Hebrón, Barcelona, Cataluny
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Del Mar, Barcelona
  - Hospital Virgen de la Arrixaca, El Palmar
  - Hospital Univ. Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Clínica Universidad de Navarra, Madrid
  - C.H. de Navarra, Pamplona
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora de Valme, Seville
  - Hospital Universitario Virgen De La Macarena, Seville
- Taiwan (5):
  - Buddihist Tzu Chi Medical Foundation- Hualien Tzu Chi Hospital, Hualien City
  - Chang Gung Medical Foundation - Kaohsiung Chang Gung Memorial Hospital - Hemato-Oncology, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (5):
  - Ankara University Medical Faculty - Hematology, Ankara
  - Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research, Ankara
  - Gazi University Medical Faculty, Ankara
  - Medipol Bagcilar Mega Hospital, Istanbul
  - Ondokuz Mayis University Medical Faculty - Hematology, Samsun
- United Kingdom (7):
  - Western General Hospital - Haematology, Edinburgh, Edinburgh, City of
  - Imperial College Healthcare NHS Trust - Hammersmith Hospital, London, London City
  - St Bartholomew's Hospital Barts Health NHS Trust, London, London, City of
  - The Clatterbridge Cancer Centre NHS Foundation Trust - Clatterbridge Cancer Centre, Bebington
  - Royal Cornwall Hospitals NHS Trust - Royal Cornwall Hospital, Cornwell
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Northwick Park Hospital Middlesex, United Kindgom, HA1 3UJ, Middlesex

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/

REFERENCES:
- [Derived] Cao J, Chen G, Qiu L, Zhang L, Jiang M, Cheng Y, Zhang Q, Liu L, Li P, Shuang Y, Wang H, Xue H, Wu H, Zheng M, Zhou K, Li Z, Jing H, Yang W, Zhu Z, Li W, Wangwu J, Huang H, Jia Q, Chen D, Fan S, Shi MM, Su W. Efficacy and safety of tazemetostat, an EZH2 inhibitor, in Chinese patients with relapsed/refractory follicular lymphoma: a multicentre, single-arm, phase 2 study. EClinicalMedicine. 2025 Aug 18;87:103399. doi: 10.1016/j.eclinm.2025.103399. eCollection 2025 Sep. PMID 40896460